CLINICAL TRIAL: NCT03745963
Title: iCAP Mini - The Influence of Skin-to-skin Contact on Cortical Activity During Painful Procedures on Preterm Infants in the Neonatal Intensive Care Unit: A Randomized Control Trial
Brief Title: The Influence of Skin-to-skin Contact on Cortical Activity During Painful Procedures on Preterm Infants in the NICU
Acronym: iCAPmini
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Principal Investigator, Marsha Campbell-Yeo, Associate Professor Dalhousie University School of Nursing, Faculty of Health, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IWKHealthC 1023060
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pain, Acute; Infant, Newborn; Electroencephalography
Keywords: Neonate; Pain; Sucrose; Skin-to-skin contact; EEG; Assessment; RCT; Bio behavioural
MeSH Terms: conditions — Acute Pain; Pain | interventions — Sucrose; Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two research assistants (RA1, RA2) who are blinded to the intervention condition will be hired to complete facial coding and calculation of infant PIPP-R scores. Each research assistant will only code data for preterm infants in the skin to skin condition (RA1) or the sucrose condition (RA2) and will not be aware of whether they are watching preterm infant responses to noxious or non-noxious stimulation. To minimize observer bias, research assistants will not be informed of the study design, will not be permitted to attend data collection sessions, and will not share datasets or communicate with the other research assistant regarding the study. During data collection, up close video recording of only the preterm infants face will be completed to attempt to keep coders blind to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Skin-to-skin contact (Experimental): Infants will be placed in full ventral skin-to-skin with their mother at least fifteen minutes prior to heel lance to allow time to settle and recover following transfer. Positioning will be determined based on individual maternal preference in order to optimize comfort as well as facilitate ease of access to the infant's foot for blood collection, while also attempting to minimize disruption of continuous EEG, heart rate, oxygen saturation, and video recording. Skin to skin contact will continue until the procedure is completed.
  In addition, infants will be offered non-nutritive sucking using a gloved finger or pacifier (based on parental preference) during SSC. Whether infants are actively sucking during the procedure will be recorded by the research coordinator.
  Interventions: Behavioral: Skin-to-skin contact
- 24% Oral sucrose (Active Comparator): Infants will be placed in a cot or in an incubator, depending on their gestational age, for the duration of the blood collection. Administration of 0.12mls (0.04mls per drop) of 24 percent oral sucrose will occur two minutes prior to the heel lance.
  The infants will be offered non-nutritive sucking using a gloved finger or pacifier (based on parental preference) immediately following administration of the complete 24 percent oral sucrose dose. Whether infants are actively sucking during the procedure will be recorded by the research coordinator.
  Interventions: Drug: 24% oral sucrose

INTERVENTIONS:
Behavioral: Skin-to-skin contact — Infants allocated to the SSC arm will be placed in upright, ventral SSC position (holding of a diaper clad baby on the bare chest of a mother) for a minimum of 15 minutes prior to data collection.
  Other Names: Kangaroo care (maternal)
  Arms: Skin-to-skin contact
Drug: 24% oral sucrose — Administration of 24 percent oral sucrose will occur two minutes prior to the heel lance.
  Other Names: sweet taste
  Arms: 24% Oral sucrose

SUMMARY:
The aim of this study is to examine the effect of SSC compared to sucrose on pain induced activity in the preterm infant brain using: a) series of low intensity experimental stimuli (PinPrick);and b) medically required heel lance. Secondary objectives include determining: a) differences between behavioral pain response and pain response during heel lance; and b) rate of adverse events across groups.

DETAILED DESCRIPTION:
Hospitalized preterm infants undergo an average of 12 painful procedures daily, with less than half receiving pain relief. Poorly treated early pain can have long lasting negative effects that impact later learning, development, and reaction to future pain, stress, and emotional experiences. While sweet tasting solution (sucrose) is considered the standard of care for reducing behavioral responses to acute procedural pain in preterm infants, some evidence that sucrose may not similarly reduce pain related brain activity raises concerns regarding the degree of pain relieving effect. This concern is especially relevant as the use of sucrose to manage repeated acute pain has not been found to prevent heightened later pain associated with this exposure. Strong evidence suggests that maternal infant skin-to-skin contact (SSC) is effective in reducing behavioral responses to pain. Given the multi-sensory benefits of SSC, it is highly likely that SSC provided during pain in early life may reduce pain induced brain activity.

Infants ( n=126) (32 to 36 completed weeks gestational age) admitted to the Neonatal Intensive Care Unit, and their mothers within the first seven days of age will be randomly assigned to receive: i) SSC or ii) 24 % oral sucrose. Each baby will receive both the PinPrick and heel lance, following a no treatment baseline period. The primary outcome is pain related brain activity measured using an electroencephalogram (EEG) pain-specific event-related potential. Secondary outcomes include pain intensity measured using a behavioural infant pain assessment tool (Premature Infant Pain Profile-Revised) and rate of adverse events.

This will be the first study to examine the effect of SSC on pain induced brain activity in the preterm infant brain during experimental and clinical pain stimuli, measured using EEG. Given the negative neurodevelopmental outcomes associated with unmanaged pain, it is imperative that preterm infants receive the most effective pain relieving treatments to improve their health outcomes.

ELIGIBILITY:
Inclusion criteria:

* stable neonates delivered between 32 and 36 completed weeks Gestational age (GA) at birth (Determination of stability will be made in consultation with the attending neonatal staff)
* admitted to NICU
* parents are able to read and write English
* will be approached for inclusion within the first seven days following birth

Exclusion criteria:

* major congenital anomalies
* receiving or received opioids in 24 hours preceding heel lance
* immediate post operative period (<72 hours) following surgery
* history of hypoxic ischemic encephalopathy requiring cooling
* contraindication for sucrose administration (e.g., unable to swallow, paralysis)

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain-specific event related potential | Isolated within the one-minute window post-procedure at lead CZ
  The primary outcome measure will be pain-specific brain activity measured using a dense array neonatal electroencephalogram (EEG) recording that is time-locked to a medically required heel lance. Infant EEG activity will be recorded from a HydroCel Geodesic Sensor Net positioned according to the modified international 10/20 electrode placement system on a 128 Channel Geodesic EEG SystemTM 400 MR series (Electrical Geodesics Incorporated, Eugene, Oregon, USA). Pain-specific event related potentials will specifically be examined and isolated at electrode sites Cz, as previous research has reported pain-specific activity at this site in both infants and adults.

SECONDARY OUTCOMES:
Premature Infant Pain Profile-Revised | Composite pain scores with be averaged over 30 second epochs and reported at 30, 60, 90, 120 seconds post heel lance
  The PIPP-R, which has been revised from the original PIPP developed 14 years ago, is a 7-indicator composite pain measure consisting of 3 behavioural (facial actions: brow bulge, eye squeeze, and naso-labial furrow), 2 physiological (heart rate, oxygen saturation) and 2 contextual (gestational age, behavioural state) indicators of acute pain. A numerical score ranging from 0 - 3 is assigned to each indicator for a maximum score of 18 reflecting the worst possible pain in infants born at greater than 36 weeks' gestational age. A score of 6 or less is considered to indicate minimal or no pain, a score of 6 to 12 indicates mild or moderate pain, and a score of 12 or greater indicates moderate to severe pain.
Recovery | The point at which the preterm infant's heart rate reaches baseline levels and is sustained for no less than five to seven beats following the heel lance, time will vary across patients but will be anticipated to be no longer than 5 minutes
  Time to recovery will be considered the amount of time in seconds that elapses until the infant's heart rate returns to baseline average values. The point at which the infant's heart rate reaches baseline levels and is sustained for no less than five to seven beats following the heel lance will indicate recovery.
Maternal acceptability: questionnaire | Immediately post-procedure
  Mothers will be asked to complete an open-ended questionnaire with 3-5 questions (depending on assigned condition) following completion of the study procedures. This questionnaire will focus on assessing maternal acceptability of the use of the assigned skin to skin contact or sweet taste intervention as well as the use of neurocognitive imaging technology to measure newborn pain responding in the neonatal period.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha L Campbell-Yeo, PhD NNP, Principal Investigator — School of Nursing, Faculty of Health, Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campbell-Yeo M, Benoit B, Newman A, Johnston C, Bardouille T, Stevens B, Jiang A. The influence of skin-to-skin contact on Cortical Activity during Painful procedures in preterm infants in the neonatal intensive care unit (iCAP mini): study protocol for a randomized control trial. Trials. 2022 Jun 20;23(1):512. doi: 10.1186/s13063-022-06424-4. PMID 35725632